CLINICAL TRIAL: NCT05178368
Title: Impact of Early Valve Replacement on Myocardial Scar in Asymptomatic Aortic Stenosis: an Observational MRI Study of Randomised Cohorts
Brief Title: MRI in Randomised Cohorts of Asymptomatic AS
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 0824
Record Dates: First submitted 2021-10-08; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-11

CONDITIONS: Aortic Stenosis, Severe
Keywords: myocardial fibrosis; cardiac magnetic resonance imaging; late gadolinium enhancement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Surgical Procedures, Operative; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collection for future ethically approved studies of biomarkers associated with fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early aortic valve replacement: Asymptomatic severe aortic stenosis patients randomised to early aortic valve replacement
  Interventions: Procedure: Surgical/ Transcatheter aortic valve replacement
- Standard care: Asymptomatic severe aortic stenosis patients randomised to 'watchful waiting' until symptom onset.

INTERVENTIONS:
Procedure: Surgical/ Transcatheter aortic valve replacement — The choice of intervention will be made by the local clinical team. The timing of intervention will be determined by randomisation as part of the main EASY/EVOLVED trials
  Groups: Early aortic valve replacement

SUMMARY:
Aortic stenosis is narrowing of the aortic valve, and is the commonest type of valve disease requiring surgery. Current guidelines recommend waiting till patients develop symptoms (chest pain, breathlessness and dizzy spells/fainting) before possible open heart surgery to replace the valve is offered. However, studies using detailed 'MRI' scanning of the heart have shown that up to half of the patients already have 'scarring' in the heart by the time symptoms develop. Furthermore, scarring is not fully reversed even after surgery and is associated with worse outcome. This suggests that some patients are being offered treatment too late. Two randomised trials in the UK (EASY AS and EVOLVED) are currently investigating if valve replacement before symptoms will result in better survival. The aim of this study is to compare the effect of early valve replacement versus waiting for symptoms, on the amount of scarring in the heart. The investigators want to know if early treatment leads to less overall scarring at the end, and leads to better quality of life and recovery after surgery. The investigators will invite participants of the EASY AS and EVOLVED trials to have 1-2 MRI heart scans: at recruitment and 3 years after being randomly allocated to early aortic valve replacement vs 'watchful waiting'. The investigators will also assess the impact of the two treatment approaches on quality of life, disability-free survival (using questionnaires) and recovery after surgery. The results from this project will increase understanding of the results of the main trials, and lead to improved selection of patients with aortic stenosis who are likely to benefit from early surgery.

DETAILED DESCRIPTION:
Ongoing randomised control trials (RCT) are testing the strategy of early AVR in asymptomatic severe AS ('The Early surgery in severe ASYmptomatic Aortic Stenosis': EASY-AS and 'Early Valve Replacement guided by Biomarkers of Left Ventricular Decompensation in Asymptomatic Patients with Severe Aortic Stenosis': EVOLVED), and if positive, have the potential to shift the timing of intervention to earlier disease. With TAVR recently being shown to be non-inferior to SAVR in low risk, mostly symptomatic patients, this also has the potential to be extended to asymptomatic patients.

MRI studies have shown that up to 50% of those with asymptomatic AS already have scarring (LGE), which is only partially reversible even after AVE, and remains a marker of mortality. It is not known if earlier valve replacement will lead to less scar burden within the myocardium.

Patient reported outcome measures (PROM) are increasingly recognised as an important outcome measure of surgery, especially in an elderly population, for whom a significant increase in survival may be neither possible, nor sought by the patient. World Health Organisation Disability Assessment Schedule-2 (WHODAS-2) is a standardised cross-cultural measurement of health status assessing functioning and disability in major life domains, that has been shown to be a valid and reliable instrument for assessment of disability. A comprehensive formal review of PROMS instruments in patients receiving medical treatment for heart failure concluded that the Euroqol (EQ5D) and Minnesota Living with Heart Failure Questionnaire (MLHFQ) were the most appropriate to measure quality of life in this group. Euroqol is the most commonly used generic instrument in Europe, and showed improvement at 1 year post-AVR for severe AS. MLHFQ is a cardiovascular disease-specific tool that has been shown to be reliable, valid and responsive to therapeutic intervention in patients undergoing valve surgery. Understanding the effect of intervention on PROMs can aid shared decision-making and help shape future individualised recommendations.

This prospective, observational mechanistic study will maximise the opportunity offered by ongoing RCTs, to try and establish the effect of the two treatment strategies (early vs late AVR) on cardiac reverse remodelling (in particular fibrosis burden), PROMs and peri-operative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to and able to consent
2. Participant in an RCT randomising patients with asymptomatic severe AS to early AVR vs standard care
3. Severe aortic stenosis, as defined by original trial's inclusion criteria
4. Asymptomatic at the time of randomisation in the RCT
5. Willingness to have 1-2 cardiac MRI scan(s)

Exclusion Criteria:

1. Contra-indication to MRI.
2. eGFR <30.
3. Severe claustrophobia (precluding MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic severe aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Total amount of fibrosis (measured by LGE on MRI) in those randomised to early AVR vs standard care. | 3 years
  Measured by percentage of late gadolinium enhancement on MRI, between those randomised to early AVR vs standard care.

SECONDARY OUTCOMES:
Differences in patient reported outcome measures (health related quality of life) between the two groups | 3 years
  Measured using the questionnaire EuroQol- 5 (EQ-5D-5L)
  EuroQol- 5 Dimension is a standardised measure of health-related quality of life and consists of 2 pages.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Differences in patient reported outcome measures (patient perceptions of living with heart failure) between the two groups | 3 years
  Measured using the Minnesota Living with Heart Failure questionnaire (MLHF)
  Minnesota Living with Heart Failure questionnaire aids to systematically and comprehensively assess the patient's perceptions of the effects of heart failure and its treatment on his or her daily life.
  It is a 21-item paper self- administered questionnaire designed as a measure of heart failure, as indicated by its adverse effects on patients' lives. The MLHFQ quantifies a single overall score as a measure of the impact of heart failure on the patient's life.
Differences in patient reported outcome measures (in assessing functioning and disability in major life domains) between the two groups | 3 years
  Measured using the World Health Organisation Disability Assessment Schedule-2 (WHODAS-2) questionnaire
  World Health Organisation Disability Assessment Schedule-2 (WHODAS-2) is a standardised cross-cultural measurement of health status assessing functioning and disability in major life domains, that has been shown to be a valid and reliable instrument for assessment of disability. It is a 36-item measure that assesses disability in adults age 18 years and older.
Difference in peri-operative recovery between the two groups. | 30 days from date of surgery
  Days at home within 30 days of surgery
Differences in reverse remodelling (by left ventricular volume) between the two groups. | 3 years
  LV end-diastolic volume index in ml/m2
Differences in reverse remodelling (by left ventricular mass) between the two groups. | 3 years
  LV mass index in g/m2
Differences in reverse remodelling (by left ventricular mass/volume) between the two groups. | 3 years
  LV mass/volume ratio
Differences in reverse remodelling (by left ventricular ejection fraction) between the two groups. | 3 years
  LV ejection fraction in %
Differences in reverse remodelling (by myocardial perfusion reserve) between the two groups. | 3 years
  Myocardial perfusion reserve (in those having optional stress perfusion)

CONTACTS AND LOCATIONS:
Overall Officials: Anvesha Singh, Dr, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom